CLINICAL TRIAL: NCT00169728
Title: Immunogenicity of the DTaP-IPV-HBV/Hib Combination Vaccine Infanrix Hexa and the Heptavalent Pneumococcal Conjugate Vaccine Prevenar in Pediatric Recipients of Allogeneic Haematopoietic Stem Cell Transplantation
Brief Title: Vaccination of Children Following Allogeneic Stem Cell Transplantation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Heinrich-Heine University, Duesseldorf (Other)
Collaborators: Wyeth is now a wholly owned subsidiary of Pfizer (Industry); GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: IKAST-01
Record Dates: First submitted 2005-09-13; First posted 2005-09-15 (Estimated); Last update posted 2012-06-07 (Estimated); Status verified 2012-06

CONDITIONS: Allogeneic Haematopoietic Stem Cell Transplantation
Keywords: allogeneic haematopoietic stem cell transplantation; bone marrow transplantation; children; vaccination; invasive pneumococcal disease; tetanus; diphtheria; poliomyelitis; pertussis; Hepatitis B; Haemophilus influenzae type B infection
MeSH Terms: conditions — Tetanus; Diphtheria; Poliomyelitis; Whooping Cough; Hepatitis B; Haemophilus Infections | interventions — diphtheria-tetanus-acellular pertussis-inactivated poliovirus-Haemophilus influenzae b conjugate-hepatitis B vaccine; Heptavalent Pneumococcal Conjugate Vaccine

INTERVENTIONS:
Biological: DTaP-IPV-HBV/Hib combination vaccine, Infanrix hexa
Biological: heptavalent pneumococcal conjugate vaccine, Prevenar

SUMMARY:
The purpose of this study is to determine the immunogenicity and tolerability of the DTaP-IPV-HBV/Hib combination vaccine Infanrix hexa and the heptavalent pneumococcal conjugate vaccine Prevenar in pediatric recipients of allogeneic haematopoietic stem cell transplantation.

ELIGIBILITY:
Inclusion Criteria:

* pediatric recipient of allogeneic haematopoietic stem cell transplantation
* complete remission of underlying malignant disease (if applicable)
* stable haematopoietic engraftment
* Lansky-/Karnofsky-score >= 60%

Exclusion Criteria:

* primary immunodeficiency
* hepatitis B or C, HIV infection
* application of radio-/ chemotherapy following stem cell transplantation
* extended chronic graft-versus-host disease (Karnofsky-scale < 60%)
* coagulopathy
* known allergy/hypersensitivity towards ingredients of study vaccines
* seizure disorder, progressive neurologic disease

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 53 (Actual)
Dates: Start 2003-09; Primary Completion 2006-06 (Actual); Study Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
serologic response at 1 months following primary three dose vaccination series | first month

SECONDARY OUTCOMES:
serologic response at 1 months following booster immunization | first month
tolerability of primary and booster vaccination | at least monthly
identification of factors influencing immunogenicity and tolerability of study vaccines | at least monthly

CONTACTS AND LOCATIONS:
Overall Officials: Dagmar Dilloo, MD, PhD, Principal Investigator — University Hospital Duesseldorf, Department of Pediatric Oncolgy, Hematolgy and Immunology
Locations (11):
- Germany (11):
  - University Childrens Hospital, Berlin
  - University Children Hospital, Düsseldorf
  - University Children Hospital, Erlangen
  - University Children Hospital, Frankfurt
  - University Childrens Hospital, Freiburg im Breisgau
  - University Childrens Hospital, Giessen
  - University Childrens Hospital, Hamburg
  - University Childrens Hospital, Hanover
  - University Childrens Hospital, Jena
  - University Childrens Hospital, Münster
  - University Childrens Hospital, Tübingen

REFERENCES:
- [Background] Meisel R, Laws HJ, Dilloo D. Vaccination of pediatric recipients of allogeneic hematopoietic stem cell grafts using a hexavalent combination vaccine and a pneumococcal conjugate vaccine - a prospective trial of the PÄD-AG-KBT - Bone Marrow Transplantation 30(S1): S63, 2002 (abstract)
- [Background] Meisel R, Dilloo D. Pneumococcal vaccination of children after hematopoietic stem cell transplantation: timing is crucial. Clin Infect Dis. 2007 Aug 1;45(3):397-8; author reply 398-9. doi: 10.1086/518981. No abstract available. PMID 17599322
- [Background] Hilgendorf I, Freund M, Jilg W, Einsele H, Gea-Banacloche J, Greinix H, Halter J, Lawitschka A, Wolff D, Meisel R. Vaccination of allogeneic haematopoietic stem cell transplant recipients: report from the international consensus conference on clinical practice in chronic GVHD. Vaccine. 2011 Apr 5;29(16):2825-33. doi: 10.1016/j.vaccine.2011.02.018. Epub 2011 Feb 20. PMID 21345379
- [Result] Meisel R, Kuypers L, Dirksen U, Schubert R, Gruhn B, Strauss G, Beutel K, Groll AH, Duffner U, Blutters-Sawatzki R, Holter W, Feuchtinger T, Gruttner HP, Schroten H, Zielen S, Ohmann C, Laws HJ, Dilloo D; Impfung von Kindern nach allogener Stammzelltransplantation (IKAST) Study Group. Pneumococcal conjugate vaccine provides early protective antibody responses in children after related and unrelated allogeneic hematopoietic stem cell transplantation. Blood. 2007 Mar 15;109(6):2322-6. doi: 10.1182/blood-2006-06-032284. Epub 2006 Nov 7. PMID 17090650